CLINICAL TRIAL: NCT07003074
Title: A Randomized, Open, Multicenter, Parallel-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQB2102 for Injection Versus Docetaxel Plus Trastuzumab and Pertuzumab in the Treatment of Human Epidermal Growth Factor Receptor 2 (HER2) Positive Recurrent or Metastatic Breast Cancer
Brief Title: A Clinical Study of TQB2102 Versus Docetaxel Plus Trastuzumab and Pertuzumab in the Treatment of HER2 Positive Recurrent or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-III-06
Record Dates: First submitted 2025-05-21; First posted 2025-06-04 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2102 for Injection (Experimental): Administer by intravenous infusion, with a 21-day treatment cycle.
  Interventions: Drug: TQB2102 for Injection
- Docetaxel combined + Trastuzumab +Pertuzumab (Active Comparator): Docetaxel: 75mg/m2, administered once every 3 weeks, intravenous infusion for 60 minutes, for a total of 6 cycles; Trastuzumab: The initial loading dose is 8mg/kg, and 6mg/kg is administered every 3 weeks thereafter; Pertuzumab: initial loading dose of 840mg, intravenous infusion for 60 minutes; Afterwards, administer 420mg every 3 weeks. After each infusion of pertuzumab, it is recommended to observe for 30-60 minutes. After the observation, trastuzumab or chemotherapy can be continued.
  Interventions: Drug: Docetaxel combined + Trastuzumab +Pertuzumab

INTERVENTIONS:
Drug: TQB2102 for Injection — TQB2102 is a next-generation HER2 Antibody-Drug Conjugate drug proposed for patients with HER2 positive Recurrent/Metastatic Breast Cancer.
  Arms: TQB2102 for Injection
Drug: Docetaxel combined + Trastuzumab +Pertuzumab — Positive control.
  Arms: Docetaxel combined + Trastuzumab +Pertuzumab

SUMMARY:
This Phase III trial adopts a randomized, open label, positive drug control, and multicenter trial design. Subjects who meet the criteria are randomly divided into 1:1 groups and receive treatment with TQB2102 injection or docetaxel combined with trastuzumab and pertuzumab, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily enrolled in this study with good compliance
* Age: 18-75 years old; Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0-1
* HER2 positive, recurrent or metastatic invasive breast cancer confirmed by histopathology or cell pathology
* Defined hormone receptor (HR) status
* Has not received systemic anti-tumor therapy during the recurrence/metastasis stage (acceptable ≤ first-line endocrine therapy)
* If receiving (new) adjuvant therapy, it is required that the time interval between the end of systemic therapy (excluding endocrine therapy) and the discovery of recurrence/metastasis be greater than 12 months
* Have at least one measurable lesion according to RECIST 1.1 criteria;
* Good major organ function

Exclusion Criteria:

* It is known that there is spinal cord compression or active central nervous system metastasis;
* Subjects with only skin and/or brain lesions as target lesions
* Combined diseases and medical history

  1. Have had or currently have other malignant tumors within the past 5 years of randomization
  2. Unrelieved toxic reactions above Common Terminology Criteria (CTC) AE grade 1 caused by any previous treatment
  3. Received major surgical treatment, open biopsy, or significant traumatic injury within 4 weeks prior to randomization
  4. There are diseases that affect intravenous injection and venous blood collection
  5. There are congenital bleeding and coagulation disorders present
  6. An arterial/deep vein thrombosis event occurred within 6 months prior to the first administration
  7. Poor blood pressure control
  8. Suffering from significant cardiovascular disease
  9. There is an uncontrolled infection of ≥ CTC AE grade 2 within 14 days before the start of treatment
  10. History of interstitial lung disease/pneumonia (non infectious) requiring steroid medication intervention in the past
  11. Individuals with moderate to severe pulmonary dysfunction/disease within 3 months prior to the first administration
  12. Active viral hepatitis with poor control
  13. Active syphilis infected individuals in need of treatment
  14. Individuals who are preparing for or have previously undergone allogeneic bone marrow transplantation or solid organ transplantation
  15. Immunosuppressants or systemic or absorbable local hormone therapy are required to achieve immunosuppression
  16. History of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases
  17. Urine routine shows urinary protein ≥++and confirms 24-hour urinary protein quantification>1.0 g
  18. Patients with renal failure requiring hemodialysis or peritoneal dialysis
  19. Poor control of diabetes
  20. Individuals with epilepsy who require treatment
  21. Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders
* Tumor related symptoms and treatment

  1. There is a third interstitial fluid accumulation or cancerous lymphangitis that cannot be controlled by drainage or other methods
  2. History of cumulative dose exposure to anthracyclines in the past
  3. Received radiation therapy within 3 weeks prior to the start of study treatment and endocrine therapy within 2 weeks prior to the start of study treatment
  4. Traditional Chinese patent medicines and simple preparations with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions within 2 weeks before the start of the study treatment
* Research treatment related

  1. Previously received antibody conjugate therapy consisting of topoisomerase I inhibitors,;
  2. Allergic to any research drug or any ingredient or excipient in the drug;
  3. Individuals who experience severe hypersensitivity reactions after using monoclonal antibodies;
  4. Participated in other clinical trials of anti-tumor therapy within 4 weeks before the start of the research treatment.
* According to the researcher's judgment, there are situations that seriously endanger the safety of the subjects or affect their ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to approximately 30 months
  According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, the proportion of subjects whose tumors are evaluated as complete response(CR) and partial response(PR) by subcenter imaging evaluation. It is recorded from the first use of the drug to disease progression or initiation of a new anticancer treatment.
Progression-Free Survival | Up to approximately 30 months
  It refers to the time between enrollment and the occurrence of objective disease progression or death caused by various reasons (whichever occurs first).

SECONDARY OUTCOMES:
Overall Survival | Up to approximately 30 months
  It refers to the time between enrollment and death caused by various reasons.
Duration of Remission | Up to approximately 30 months
  The subjects with the best response determined according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria as complete response (CR) or partial response (PR) are defined as the period from the first recorded tumor response to the first recorded disease progression or death from any cause, whichever occurs first.
The incidence of adverse events | Up to approximately 52 months
  During the period from the signing of the informed consent form by the subjects to 28 days after the last dose of medication/initiation of new anti-tumor treatment (based on the first occurrence), the incidence of adverse events was recorded according to the common adverse event (AE) evaluation criteria of the National Cancer Institute (NCI CTC AE 5.0 version).
The severity of adverse events | Up to approximately 52 months
  During the period from the signing of the informed consent form by the subjects to 28 days after the last dose of medication/initiation of new anti-tumor treatment (based on the first occurrence), the severity of adverse events was recorded according to the common AE evaluation criteria of the National Cancer Institute (NCI CTCAE 5.0 version).
Blood concentrations of the Antibody-Drug Conjugate (ADC) drug TQB2102 | Within 1 hour prior to the start of infusion for Cycle 1, Cycle 2,,Cycle 4, Cycle 8and 15 minutes after the end of infusion for Cycle 2, Cycle 4, (21 days as a treatment cycle)
  To evaluate the pharmacokinetic (PK) profile of TQB2102 for injection in subjects with HER2 low-expressing recurrent/metastatic breast cancer.
The incidence of drug-resistant antibodies (ADA) and neutralizing antibodies (NAb) | within 60 minutes prior to the start of infusion for Cycle 1, Cycle 2,,Cycle 4, Cycle 8, Cycle16,and before administration and 28 days (± 7 days), (21 days as a treatment cycle)
  The incidence of drug-resistant antibodies (ADA) and neutralizing antibodies (NAb)
Total antibodies | Within 1 hour prior to the start of infusion for Cycle 1, Cycle 2,,Cycle 4, Cycle 8and 15 minutes after the end of infusion for Cycle 2, Cycle 4, (21 days as a treatment cycle)
  To evaluate the pharmacokinetic (PK) profile of TQB2102 for injection in subjects with HER2 low-expressing recurrent/metastatic breast cancer.
The small molecule toxin TQ22723 | Within 1 hour prior to the start of infusion for Cycle 1, Cycle 2,,Cycle 4, Cycle 8and 15 minutes after the end of infusion for Cycle 2, Cycle 4, (21 days as a treatment cycle)
  To evaluate the pharmacokinetic (PK) profile of TQB2102 for injection in subjects with HER2 low-expressing recurrent/metastatic breast cancer.

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Tiantan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Shantou Central Hospital, Shantou, Guangdong
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - The Third People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital Of Dalian University, Dalian, Liaoning
  - Liaoning Provincial Cancer Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'An Jiaoting Yniversity, Xi'an, Shaanxi
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Fudan University shanghai cancer center, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Yuncheng Central Hospital, Shanxi Province, Yuncheng, Shanxi
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang